CLINICAL TRIAL: NCT01914302
Title: Lancing Device Blood Volume Study
Brief Title: The Characterization of Blood Volumes of Commercially Available Lancing Devices
Status: Completed | Type: Observational
Sponsor: Facet Technologies (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Sponsor
Other Study IDs: FT6000682013
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Delica Lancing Device: Subjects in this group either use the Delica lancing device or a meter that requires 1.0 microliters of blood
  Interventions: Device: Delica Lancing Device
- Freestyle Flash Lancing Device: Subjects in this group either use the Flash lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Flash Lancing Device
- Easy Touch Lancing Device: Subjects in this group either use the Easy Touch lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Easy Touch Lancing Device
- Glucoject Lancing Device: Subjects in this group either use the Glucoject lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Glucoject Lancing Device
- Microlet Lancing Device: Subjects in this group either use the Microlet lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Microlet Lancing Device
- Multiclix Lancing Device: Subjects in this group either use the Multiclix lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Multiclix Lancing Device
- Fastclix Lancing Device: Subjects in this group either use the Fastclix lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Fastclix Lancing Device
- Reli-On Lancing Device: Subjects in this group either use the Reli-On lancing device or a meter that requires 0.3/0.6 microliters of blood
  Interventions: Device: Reli-On Lancing Device

INTERVENTIONS:
Device: Delica Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Delica Lancing Device
Device: Flash Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Freestyle Flash Lancing Device
Device: Easy Touch Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Easy Touch Lancing Device
Device: Glucoject Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Glucoject Lancing Device
Device: Microlet Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Microlet Lancing Device
Device: Multiclix Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Multiclix Lancing Device
Device: Fastclix Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Fastclix Lancing Device
Device: Reli-On Lancing Device — Characterize Blood Volume and Pain under normal use circumstances
  Groups: Reli-On Lancing Device

SUMMARY:
Characterize expressed blood volume ≥1μL across representative, commercially available lancing device systems using finger sticks.

DETAILED DESCRIPTION:
Primary Objective:

• Characterize expressed blood volume ≥1μL across representative, commercially available lancing device systems using finger sticks.

Secondary Objectives: the following characterizations will be performed in the data analysis within each device and across each device:

* Correlation of Subject pain response to blood volume collected;
* Proportion of Subjects that produce sufficient blood to fill a 1µl test strip;
* Proportion of Subjects that generate ≥1µl blood volume;
* Proportion of Subjects who generate multiple- times the blood volume needed to fill a 1µl test strip
* Proportion of Subjects who generate multiple- times ≥1µl of blood volume
* Proportion of Subjects that produce on average (≥1µl) of blood volume on 1st attempt
* Proportion of Subjects that produce on average (≥1µl) of blood volume on their first and second lancing attempt

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with type 1 or type 2 diabetes for one (1) or more year(s).
* Must be currently self-monitoring blood glucose levels for at least 6 months.
* Must self-test at least 2 times daily.
* Must be between the ages of 18 and 75 to participate.
* Subjects must be able to perform all tasks required in this protocol.
* Subjects must be willing to complete all study procedures.
* Subjects must be able to speak, read and understand English and understand the Informed Consent document.

Exclusion Criteria:

* Subjects with neuropathy or any other nerve damage in the hand or fingers (this will be discovered through the monofilament test)
* Subjects who are taking prescription anti-coagulants or more than one full aspirin per day during the past week or have clotting problems that may prolong bleeding (persons taking Plavix or a daily low dose aspirin will not be excluded but this will be recorded).
* Subjects taking pain relievers within 24 hours.
* Subjects with hemophilia or any other bleeding disorder.
* Subjects with infection with a blood borne pathogen (e.g., HIV, hepatitis).
* Subjects having a condition such as a cognitive disorder, which in the opinion of the Investigator would put the person at risk or seriously compromise the integrity of the study (PI will sign Case Report Form if Subject is excluded).
* Subjects working for Facet, LifeScan Inc., or a competitive company.
* Subjects with missing digits.
* Subjects who are pregnant or nursing.
* Subjects on chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with diabetes
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood Volumes measured in microliters | between 1 and 10 days after first visit
  Study subject lances assigned finger and acquires blood drop; at that time the study facilitator gathers blood in pipette and measures on scale

SECONDARY OUTCOMES:
Pain rating measure on a 0-20 Gracely Scale | between 1 and 10 days after first visit
  Subjects were asked to rate pain on Gracely scale after each lancing even on the finger

CONTACTS AND LOCATIONS:
Overall Officials: Barry Ginsberg, MD, Principal Investigator
Locations (1):
- Facet Technologies, Kennesaw, Georgia, United States